CLINICAL TRIAL: NCT03675347
Title: Incidence, Predictors and impAct on General Population of Recurrent Events After Percutaneous Coronary INterventio for ACS: the AGAIN a Multicenter Study
Brief Title: Recurrent Events After Percutaneous Coronary INterventio for ACS
Acronym: AGAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Director, A.O.U. Città della Salute e della Scienza
Other Study IDs: AGAIN
Record Dates: First submitted 2018-09-07; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: angioplasty — angioplasty

SUMMARY:
Patients undergoing PCI for ACS are exposed to a significant ischemic and bleeding risk.

The aim of our study is instead to analyze in detail the rates of recurrent events, but also their predictors and impact on outcomes, in a population of unselected real life patients treated with PCI for ACS discharged on either Clopidogrel, Prasugrel or Ticagrelor who already experienced an adverse event during the first year of follow up.

DETAILED DESCRIPTION:
Patients undergoing PCI for ACS are exposed to a significant ischemic and bleeding risk. The rate, predictors and outcomes of an adverse event in this population has been already investigated. However, to the best of our knowledge, only two papers took specifically in analysis rates of recurrence after a first event; the first is a recently published article by Giustino et al; it took in consideration recurrent events in a selected population of patients with ST-elevation Myocardial Infarction (STEMI) participating in the HORIZONS-AMI Trial, discharged on Aspirin and Clopidogrel, analyzing their incidence in the first year of follow-up. The second is a paper by Fanaroff et al which primarily focused on the factors leading to a DAPT intensification in patients with recurrent events.

The aim of our study is instead to analyze in detail the rates of recurrent events, but also their predictors and impact on outcomes, in a population of unselected real life patients treated with PCI for ACS discharged on either Clopidogrel, Prasugrel or Ticagrelor who already experienced an adverse event during the first year of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria in the present study was the occurrence of an adverse event (bleeding or ischemic) during DAPT therapy in the follow-up after PCI for ACS

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Coronary Syndrome (ACS) treated with Percutaneous Coronary Intervention (PCI) who experienced a bleeding or ischemic event during the first year of follow-up
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Rates of recurrent bleeding and ischemic events after PCI for ACS | 2018 - 2019
  Bleedings events are defined as type 2-5 according to the Bleeding Academic Research Consortium (BARC) definition. Ischemic events are defined as myocardial infarction (MI) and definite stent thrombosis (ST).

CONTACTS AND LOCATIONS:
Overall Officials: biole carloalberto, doctor, Study Chair — Molinette
Locations (1):
- San Giovanni Battista, Torino, Italy

IPD SHARING:
Plan to Share IPD: No